CLINICAL TRIAL: NCT01595555
Title: Effectiveness of an Internet-based Mindfulness Program for Stress Management
Brief Title: Effectiveness of Stress Free Now: an Internet-based Mindfulness Program for Stress Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: General Electric (Industry)
Responsible Party: Principal Investigator, Linda Libertini, Research Coordinator, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10-278
Record Dates: First submitted 2012-05-08; First posted 2012-05-10 (Estimated); Last update posted 2022-05-11 (Actual); Status verified 2022-05

CONDITIONS: Healthy Individuals With Perceived Stress
Keywords: stress; relaxation; mindfulness; web-based; online; social media; discussion board

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Wait-list control (No Intervention): Group with no intervention. Only complete questionnaires at baseline, week 8 and 12 and activity logs through the first 8 weeks
- Stress Free Now (Experimental): Participate in the 8 week online stress management program Stress Free Now. Complete questionnaires at baseline, week 8 and 12 and activity logs through the first 8 weeks
  Interventions: Behavioral: Stress Free Now
- Stress Free Now + Social Media (Experimental): Participate in the 8-week Stress Free Now program and a discussion board that provides peer and moderator support. Complete questionnaires at baseline, week 8 and 12 and activity logs through the first 8 weeks
  Interventions: Behavioral: Stress Free Now

INTERVENTIONS:
Behavioral: Stress Free Now — 8 week mindfulness online program with the following content: 8 Weekly lesson of the week (audio), 8 Weekly mindfulness practice (audio), Daily articles on concepts and information about stress, relaxation and mindfulness, Daily motivational quotes and tips, Biweekly email reminder to participate in the program.
  Arms: Stress Free Now; Stress Free Now + Social Media

SUMMARY:
This research will examine whether an Internet-based mindfulness program for stress management produced positive outcomes for participants and is technologically feasible

DETAILED DESCRIPTION:
Chronic, severe stress, a risk factor for premature aging and myocardial infarction, affects 35% of North Americans. Stress management programs, while effective, may be prohibitively resource intensive or difficult to access by broad populations.

This research is examining whether an online stress management program - Stress Free Now© (SFN) - can achieve meaningful improvements in measures of stress and wellbeing. We are also examining whether improvements in wellbeing and stress can be enhanced through an online, internet based support group which share experiences as they go through the Stress Free Now program. This program is modeled after an intensive group program, called Mindfulness Based Stress Reduction (MBSR), which has shown benefits across a broad array of medical issues in addition to more specific stress related problems.

This is a three arm randomized controlled trial which will last for 12 weeks. Participants will be randomized into one of the study arms: Non intervention Control, Stress Free Now and Stress Free Now + Message Board. We aim at enrolling 600 participants, with the expectation that 50% will complete the study (100 per group).

A series of questionnaires will be collected at baseline, at the end of the 8-week program and at follow up at week 12. Outcome measured are stress, mindfulness, vitality, physical, social and emotional health, transcendence and self-acceptance. We will also ask participants to complete a weekly log to measure program adherence and usage.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Sign-up for SFN (if in one of the intervention groups)
* Agree to participate in the research
* Have regular access to the internet

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 684 (Actual)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Effect of SFN on stress | End of intervention at week 8
  Assess whether SFN reduces stress as measured by the Perceived Stress Scale (PSS)
Effect of SFN on mindfulness | End of intervention at week 8
  Assess whether SFN improves mindfulness as measured by the Mindfulness Attention Awareness Scale (MAAS)
Effect of SFN on self acceptance | End of intervention at week 8
  Assess whether SFN improves self-acceptance as measured by the Psychological Well-being - Self-Acceptance Subscale (PWb-SA)
Effect of SFN on vitality | End of intervention at week 8
  Assess whether SFN improves vitality as measured by the Subjective Vitality Scale (SVS)
Effect of SFN on spirituality | End of intervention at week 8
  Assess whether SFN improves transcendence as measured by the Adult Self-Transcendence Inventory (ASTI)

SECONDARY OUTCOMES:
SFN effect on physical and mental health | End of intervention at week 8
  Assess whether psycho-emotional improvement was accompanied with physical and mental health improvement as measured by SF36
Effect maintained at week 12 follow up | Week 12
  To assess whether outcome improvements are maintained at week 12
Assess whether adding Social Media to SFN improves engagement and outcome | Week 8 and 12
  To explore whether adding a message board component would enhance the effectiveness and experience of the program for participants
Assess program engagement and adherence | Through the 8-week program
  Assess program engagement and adherence by collecting Stress Free Now and Social Media self report weekly practice data and Website usage

CONTACTS AND LOCATIONS:
Overall Officials: Didier Allexandre, Ph.D., Principal Investigator — The Cleveland Clinic; Tom Morledge, M.D., Principal Investigator — Revati Wellness
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

REFERENCES:
- See also: Link to the Stress Free Now online program — http://www.clevelandclinicwellness.com/programs/Pages/StressFreeNow.aspx